CLINICAL TRIAL: NCT02752217
Title: Effectiveness of Inspiratory Muscle Training With Antihypertensive Breathing Technique on Lung and Exercise Capacity in Elderly With Isolated Systolic Hypertension
Brief Title: Effectiveness of Inspiratory Muscle Training With Slow Breathing in Elderly With ISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Phailin Tongdee, Effectiveness of inspiratory muscle training with antihypertensive breathing technique on lung and exercise capacity in elderly with isolated systolic hypertension, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE 581469
Record Dates: First submitted 2016-04-07; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Training (IMT) (Experimental): Subjects in the inspiratory muscle training (IMT) group will perform loaded deep breathing exercise at 6 breaths/min using BreatheMaxยฎ device. The IMT protocol at 6 breathing rate (inspiratory time = 4 seconds and expiratory time = 6 seconds) with load at 25 percent of MIP for eighth weeks.
  The pressure will be control by pressure manometer and duty cycle are control by subjects count duration for inspiration and expiration during training. The program will perform at home for 10 breaths/min/set, 6 sets/day with at least 1 minutes rest between sessions, 7 days/week for 8 weeks
  Interventions: Other: Inspiratory Muscle Training
- Control (Placebo Comparator): Subjects in the control (CON) group will perform breathing exercise with inspiratory load at 2 cmH2O at 6 breathing rate using one BreatheMAXยฎ device. The pressure will be control by pressure manometer and duty cycle are control by subjects count duration for inspiration and expiration during training. The program will perform at home for 10 breaths/min/set, 6 sets/day with at least 1 minutes rest between sessions, 7 days/week for 8 weeks
  Interventions: Other: Control

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training at 25%MIP with Slow breathing at 6 breath per min with BreatheMAX device for 8 weeks at home
  Arms: Inspiratory Muscle Training (IMT)
Other: Control — Inspiratory muscle training at 2 cmH2O with Slow breathing at 6 breath per min with BreatheMAX device for 8 weeks at home
  Arms: Control

SUMMARY:
Study the effects of inspiratory muscle training at Low load of 25 %Maximal inspiratory pressure with slow breathing rate at 6 breaths/min on inspiratory muscle strength, lung function, chest wall expansion, abdominal expansion, exercise capacity and blood pressure in elderly with Isolated systolic hypertension.

DETAILED DESCRIPTION:
Study the effects of inspiratory muscle training at Low load of 25 % Maximal inspiratory pressure with slow breathing rate at 6 breaths/min with BreatheMAXยฎdevice for 8 weeks at home on inspiratory muscle strength, lung function (slow vital capacity, inspiratory capacity), chest wall expansion, abdominal expansion, exercise capacity by arm ergometry and blood pressure in elderly with Isolated systolic hypertension. who have age 60-80 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 60 to 80 years of age with an essential isolated systolic hypertension stage I II based on recommendation of JNC VII from primary care units in community and the Outpatient Department of Srinakarind hospital in Khon Kaen province Thailand
2. Good communication and co operation
3. Independent physical activity
4. Stable controlled hypertension

Exclusion Criteria:

1. Essential isolated systolic hypertension stage III or secondary hypertension
2. History of heart disease such as coronary artery disease myocardial infarction
3. History of respiratory disease such as asthma chronic bronchitis
4. History of neuromuscular disease such as muscle weakness cerebrovascular disease
5. History of renal disease
6. Exercise limited by pain

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Maximal inspiratory pressure (MIP) | Baseline and at 8 weeks
  MIP will be measure by Mouth pressure meter (Micro RPM, Micro Medical, Inc., Chatham Maritime, Kent)

SECONDARY OUTCOMES:
Lung capacity | Baseline and at 8 weeks
  Lung capacity consists of slow vital capacity (SVC), inspiratory capacity (IC). SVC and IC will be measure by a portable computerized spirometer (KoKo spirometer)
Exercise capacity | Baseline and at 8 weeks
  Exercise capacity by Arm ergometer consists of exercise times, rating of perceived breathlessness (RPB) will examined by Borg scale
Chest wall expansion and abdominal expansion | Baseline and at 8 weeks
  chest wall expansion and abdominal expansion measured at xiphoid process level and middle between the ambrical and xiphiod process level by use a flexible measuring tape (cm)
Blood pressure (BP) | Baseline and at 8 weeks
  Blood pressure (BP) at home measured by digital bedside monitor. Accordingly follow ACMS recommended. And BP at laboratory test measured by Bedside monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Phailin Tongdee, Master, Principal Investigator — Faculty of Associated Medical Sciences.
Locations (1):
- Faculty of Associated Medical Sciences, Na Muang, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jones CU, Sangthong B, Pachirat O. An inspiratory load enhances the antihypertensive effects of home-based training with slow deep breathing: a randomised trial. J Physiother. 2010;56(3):179-86. doi: 10.1016/s1836-9553(10)70023-0. PMID 20795924
- [Derived] Ublosakka-Jones C, Tongdee P, Pachirat O, Jones DA. Slow loaded breathing training improves blood pressure, lung capacity and arm exercise endurance for older people with treated and stable isolated systolic hypertension. Exp Gerontol. 2018 Jul 15;108:48-53. doi: 10.1016/j.exger.2018.03.023. Epub 2018 Mar 28. PMID 29604403
- See also: An inspiratory load enhances the antihypertensive effects of home-based training with slow deep breathing: a randomised trial. — http://www.ncbi.nlm.nih.gov/pubmed/?term=An+inspiratory+load+enhances+the+antihypertensive++effects+of+home-based+training+with+slow+deep+breathing%3A+a+randomised+trial.